CLINICAL TRIAL: NCT02381769
Title: THE IMMUNOLOGICAL EFFECTS AND METABOLIC TOLERANCE OF LIPID INFUSION IN PATIENTS WITH CIRRHOSIS.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: ILBS-lipid infusion-01
Record Dates: First submitted 2015-02-23; First posted 2015-03-06 (Estimated); Last update posted 2016-09-12 (Estimated); Status verified 2014-12

CONDITIONS: Alcoholic Liver Disease
MeSH Terms: conditions — Liver Diseases, Alcoholic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Parenteral Nutrition (Experimental): Soybean based lipid emulsion
  Interventions: Dietary Supplement: Soybean based lipid emulsion

INTERVENTIONS:
Dietary Supplement: Soybean based lipid emulsion

SUMMARY:
The study will be an experimental pre-post trial in which patients with ethanol related liver disease (both severe alcoholic hepatitis and decompensated ) admitted in our institute from Jun 2013-Dec 2014 will be enrolled in the study. Those on ryle's tube feeding would receive polymeric blenderized kitchen based liquid diet while those tolerating orally would receive soft/ solid diet as tolerated as per requirement. All the patients would receive same amount of calories i.e., 30-35 kcal/kg ideal body weight/ day and 1-1.2 gm/kg protein. 35-40% of non protein calorie would be provided as fats and rest of the calories will be provided as carbohydrates. All patients will be transfused 250ml of 20% intra lipid per day for 3 consecutive days, over and above the feed provided to them to be taken enterally (orally or through Ryle's Tube). Patients will undergo tests prior to infusion and 72 hours after infusion.

ELIGIBILITY:
'Inclusion Criteria:

* Subjects aged ≥ 18 years.
* Patients with alcohol related liver disease (severe alcoholic hepatitis and decompensated cirrhosis)
* Patients tolerating enteral nutrition.

Exclusion Criteria:

* Active ongoing Gastrointestinal bleed.
* Unresolved sepsis
* Allergy to soya oil, eggs, peanuts or other ingredients of intralipid.
* Co-morbidities like Diabetes mellitus, hyperlipidemia, Coronary Artery Disease (CAD) and hypothyroidism.
* Renal failure (S.creatinine > 1.5mg %)
* Pregnancy
* Patients on high inotropic support (requiring more than 1 inotropic support)
* Refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2013-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Effect of intravenous lipid on monocytes counts. | 3 days
Effect of intravenous lipid on neutrophils counts. | 3 days
Effect of intravenous lipid on macrophages count. | 3 days

SECONDARY OUTCOMES:
Influence of lipid infusion on TEG (Thromboelastography) | 3 days
Influence of lipid infusion on TNF-α (Tumor Necrosis Factor). | 3 days
Influence of lipid infusion on interleukin levels (IL-6, IL-10). | 3 days
Influence of lipid infusion on PT/INR | 3 days
Influence of lipid infusion on PTT. | 3 days
Influence of lipid infusion on liver parameters. | 3 days
Influence of lipid infusion on arterial ammonia. | 3 days
Influence of lipid infusion on renal parameters. | 3 days

OTHER OUTCOMES:
Influence of lipid infusion on nitrogen balance | 3 days
  nitrogen balance would be calculated by 24 hours urinary blood urea nitrogen estimation.
Metabolic tolerance of lipid infusion. | 3 days
  Metabolic tolerance would be assessed by effect on serum triglycerides level ,serum free fatty acid level,arterial lactate level.
Effect of lipid infusion on Oxidative stress. | 3 days
  Oxidative stress would be determine by using urinary isoprostane test.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India